CLINICAL TRIAL: NCT02108015
Title: Evaluation of a Novel Positron Emission Tomography (PET Radiotracer for TARP Gamma-8
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140068; 14-M-0068
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2014-09-05

CONDITIONS: Healthy Volunteers
Keywords: Transmembrane AMPA Receptor Regulatory Protein; Glutamate Receptors; Healthy Volunteers
MeSH Terms: interventions — Neuroimaging; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Blood Specimen Collection

INTERVENTIONS:
Procedure: Brain Imaging (PET)
Procedure: Aterial Line
Procedure: Blood Sampling

SUMMARY:
Objective

Ionotropic glutamate receptors are ligand-gated ion channels responsible for most of the excitatory neurotransmission in the mammalian central nervous system (CNS). Based on pharmacology, they have been grouped into three subtypes-NMDA, AMPA and kainate. In recent years it has become apparent that the receptors do not function alone, but in the company of auxiliary proteins that regulate their activity [1]. Some of these have been shown to modulate AMPA receptor trafficking, gating and pharmacology and are classified as transmembrane AMPA receptor regulatory proteins, or TARPs ( >=-2, >=-3, >=-4, >=-5, >=-7, and >=-8). Genetic data indicate a possible role of TARPs in schizophrenia, depression, epilepsy, neuropathic pain, and bipolar disorder [1]. In a preclinical collaboration with Eli Lilly, we developed a promising radioligand, 18F-TARP252 to image TARP >=-8 using positron emission tomography (PET).

This protocol covers three phases:

* Phase 1: kinetic brain imaging to quantify TARP >=-8 in brain relative to concurrent measurement of the parent radioligand in arterial plasma;
* Phase 2: if 18F-TARP252 is successful in Phase 1, we will estimate the radiation-absorbed doses by performing whole body imaging;
* Phase 3: test-retest analysis of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma.

Study Population

Healthy adult female and male volunteers (n=22, ages 18 - 55) will undergo brain imaging. An additional eight healthy volunteers will undergo whole body dosimetry analysis.

Design

For quantification of TARP >=-8, 22 healthy controls will have brain PET imaging using 18F-TARP252 and an arterial line. Some of them will have a test-retest scan. Eight additional subjects will have a whole body PET scan for dosimetry. For dosimetry, no arterial line will be used.

Outcome Measures

To assess quantitation of TARP >=-8 with 18F-TARP252, we will primarily use two outcome measures: the identifiability and time stability of distribution volume calculated with compartmental modeling. In test-retest study, we will calculate the retest variability. We will assess whole-body biodistribution and dosimetry of 18F-TARP252 by calculating doses to organs and effective dose to the body.

DETAILED DESCRIPTION:
Objective

Ionotropic glutamate receptors are ligand-gated ion channels responsible for most of the excitatory neurotransmission in the mammalian central nervous system (CNS). Based on pharmacology, they have been grouped into three subtypes-NMDA, AMPA and kainate. In recent years it has become apparent that the receptors do not function alone, but in the company of auxiliary proteins that regulate their activity [1]. Some of these have been shown to modulate AMPA receptor trafficking, gating and pharmacology and are classified as transmembrane AMPA receptor regulatory proteins, or TARPs ( >=-2, >=-3, >=-4, >=-5, >=-7, and >=-8). Genetic data indicate a possible role of TARPs in schizophrenia, depression, epilepsy, neuropathic pain, and bipolar disorder [1]. In a preclinical collaboration with Eli Lilly, we developed a promising radioligand, 18F-TARP252 to image TARP >=-8 using positron emission tomography (PET).

This protocol covers three phases:

* Phase 1: kinetic brain imaging to quantify TARP >=-8 in brain relative to concurrent measurement of the parent radioligand in arterial plasma;
* Phase 2: if 18F-TARP252 is successful in Phase 1, we will estimate the radiation-absorbed doses by performing whole body imaging;
* Phase 3: test-retest analysis of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma.

Study Population

Healthy adult female and male volunteers (n=22, ages 18 - 55) will undergo brain imaging. An additional eight healthy volunteers will undergo whole body dosimetry analysis.

Design

For quantification of TARP >=-8, 22 healthy controls will have brain PET imaging using 18F-TARP252 and an arterial line. Some of them will have a test-retest scan. Eight additional subjects will have a whole body PET scan for dosimetry. For dosimetry, no arterial line will be used.

Outcome Measures

To assess quantitation of TARP >=-8 with 18F-TARP252, we will primarily use two outcome measures: the identifiability and time stability of distribution volume calculated with compartmental modeling. In test-retest study, we will calculate the retest variability. We will assess whole-body biodistribution and dosimetry of 18F-TARP252 by calculating doses to organs and effective dose to the body.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 - 55 (including 18 and 55).
* Able to give written informed consent.
* Healthy
* Enrolled in 01-M-0254

EXCLUSION CRITERIA:

* Any current Axis I diagnosis.
* Clinically significant laboratory abnormalities.
* Positive HIV test.
* Unable to have an MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* Recent exposure to radiation related to research (i.e. PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* Drug/alcohol abuse or dependence

Exclusion criteria for the dosimetry subjects are the same as reported above, with the exception of MRI contraindications, because an MRI will not be performed in these subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03-05; Primary Completion 2014-09-05 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Binding of 18F-TARP252 in brain | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kato AS, Gill MB, Yu H, Nisenbaum ES, Bredt DS. TARPs differentially decorate AMPA receptors to specify neuropharmacology. Trends Neurosci. 2010 May;33(5):241-8. doi: 10.1016/j.tins.2010.02.004. Epub 2010 Mar 8. PMID 20219255
- [Background] Letts VA, Felix R, Biddlecome GH, Arikkath J, Mahaffey CL, Valenzuela A, Bartlett FS 2nd, Mori Y, Campbell KP, Frankel WN. The mouse stargazer gene encodes a neuronal Ca2+-channel gamma subunit. Nat Genet. 1998 Aug;19(4):340-7. doi: 10.1038/1228. PMID 9697694
- [Background] Chen L, Chetkovich DM, Petralia RS, Sweeney NT, Kawasaki Y, Wenthold RJ, Bredt DS, Nicoll RA. Stargazin regulates synaptic targeting of AMPA receptors by two distinct mechanisms. Nature. 2000 Dec 21-28;408(6815):936-43. doi: 10.1038/35050030. PMID 11140673